CLINICAL TRIAL: NCT03717324
Title: Identifying Improvements in an Emergency Department Elder Friendly Area Based on Patient Experience (EDEFA_TheirVoice Project)
Brief Title: Identifying Improvements in an ED Elder Friendly Area Based on Patient Experience (EDEFA_TheirVoice Project)
Acronym: TheirVoice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IIBSP-EXP-2018-80
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Emergencies; Aging
Keywords: Emergency Department; Geriatrics; Frailty
MeSH Terms: conditions — Emergencies; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First evaluation group (survey_1): Patients/caregivers attended in the Emergency Department Elder Friendly Area (EFA)
- Co-creation group: Patients/caregivers attended in the Emergency Department Elder Friendly Area (EFA) who want to participate in the co-creation workshop
  Interventions: Other: Procedure created in co-creation group
- Second evaluation group (survey_2): Patients/caregivers attended in the Emergency Department Elder Friendly Area (EFA), after improvements are made
  Interventions: Other: Procedure created in co-creation group

INTERVENTIONS:
Other: Procedure created in co-creation group — Interventions will be those obtained from the co-creation workshop with patients
  Groups: Co-creation group; Second evaluation group (survey_2)

SUMMARY:
Analyze patient experience of elders admitted to the Emergency Department Elder Friendly Area (EFA) and determine possible improvement options and potential solutions.

The project will use a creative problem-solving methodology (Design Thinking) to analyze the care process based on the experience of Elder Friendly Area (EFA) users and their families

DETAILED DESCRIPTION:
Method: This is a qualitative and quantitative evaluation project. The project will use a creative problem-solving methodology (Design Thinking) to analyze the care process based on the experience of Elder Friendly Area (EFA) users and their families. Design Thinking is a creativity and innovation methodology that compiles tools based on design principles for problem solving. It is characterized by having the ability to mix convergent and divergent thinking, reconciling rational and intuitive thinking. This methodology consists of 4 phases: Mapping, Exploring, Building and Testing. In each of them, the tools and techniques help us to observe, get involved and immerse ourselves in the patient's ecosystem, with the aim of designing a solution WITH the user and not just FOR him. Consequently, the error is reduced and the modifications and improvements of our projects are speeded up.

Patients: Patients/caregivers attended in the Emergency Department's EFA will participate . In the first fieldwork, 50-60 patients will participate, conducting a self-completed interview (prior informed consent, 10 minutes long).

In the qualitative research phase, 5-10 patients/caregivers conduct a 30-minute interview with the Design Thinking professional. The co-creation workshop lasts a couple of hours and 5 to 10 patients/caregivers will participate. In the second fieldwork another 50-60 patients will participate. In total, between 110 and 140 patients will be enrolled.

Ethics: Patients/caregivers will be provided with a patient information sheet and informed consent prior to participation. Patient experience data will be collected by Design Thinking professional on an anonymous basis and will always be handled on an aggregate basis.

Funding: The project will be developed in collaboration with Merck Sharp & Dohme Spain, with which there is an agreement signed (Fundació de Gestió HSCSP - MSD). For the correct development of it, MSD has hired a company expert in the development of this type of dynamics (Thinkers&Co) which will participate actively in all meetings and workshops and will be responsible for collecting the opinion of the patient anonymously and manage this information in an aggregate way, always with the intention of identifying the points of improvement on which later health professionals will work with the methodology described. However, no monetary payment will be made to the hospital, to the emergency department or to the professionals involved. The collaboration of MSD and Thinkers&Co will not affect the independent nature of the project.

ELIGIBILITY:
Inclusion Criteria:

* All patients attended in elder friendly area who agree to participate and their caregivers

Exclusion Criteria:

* None

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients attended in elder friendly area who agree to participate and their caregivers. All them are old frail people.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2018-11-22 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative improvement in the satisfaction survey | 1 month
  A quantitative increase in the satisfaction survey obtained after the improvement implemented after the co-creation workshop.

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Puig, Principal Investigator — Hospital de la Santa Creu i Sant Pau, Emergency Department
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided